CLINICAL TRIAL: NCT04638231
Title: Supportive Text Messaging Versus Supportive E-mail Messaging for Patients with Major Depressive Disorder - a Non-Inferiority Randomized Trial
Brief Title: Supportive Text Messaging Versus Supportive E-mail Messaging for Patients with Major Depressive Disorder
Acronym: STEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00105429
Record Dates: First submitted 2020-11-07; First posted 2020-11-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-03

CONDITIONS: Major Depressive Disorder
Keywords: Email messaging; Text messaging; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: This is a two-arm randomized non-inferiority pilot trial in which patients with MDD receiving usual care are randomized to receive either daily supportive email messaging or daily supportive text messaging of the same content.
Who Masked: Investigator
Masking Description: We will use block randomization with a series of computer-generated random numbers to ensure balance (1:1) between the two treatment groups. The randomisation codes will be transmitted by an independent statistician via text message directly to the blinded researcher's password-protected phone line with a secure online backup
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Text Message Group (Active Comparator): This group will receive daily supportive messages through Short Messaging Service (SMS) on their mobile phones in addition to standard care
  Interventions: Other: Supportive messages
- Email Message Group (Experimental): This group will receive same supportive message as the Text Message group but through their email addresses, in addition to receiving standard care
  Interventions: Other: Supportive messages

INTERVENTIONS:
Other: Supportive messages — Daily supportive messages via SMS or email

SUMMARY:
Background: In 2012, over 3.2 million Canadians over 15 (11.3%) years reported symptoms of major depressive disorder (MDD), and barriers such as lack of readily available care system, stigma and affordability of health care services were reported by millions of Canadians who expressed they had unmet or partially met mental health care needs. There is the need to develop innovative psychological interventions which are not human resource intensive, are easily accessible, cost-effective, are geographic location independent, scalable, and can be offered to thousands of people simultaneously. Supportive text messaging has been proven in clinical trials to be effective in alleviating depression symptoms but are limited in their ability support those without active cell phones.

Objective: The objective of this study is to evaluate the feasibility, comparative effectiveness and user satisfaction with daily supportive e-mail messaging as an intervention to treat patients with MDD when compared to daily supportive text messaging.

Method: In this innovative two-arm randomized non-inferiority pilot trial, patients with MDD receiving usual care would be randomized to receive either daily supportive email messaging or daily supportive text messaging of the same content for six months. The Patient Health Questionnaire (PHQ)-9 scale will be utilized to record depression symptom scores, the Generalized Anxiety Disorder (GAD)-7 scale would be used to record the anxiety symptoms and quality of life will be measured using the WHO (Five) Well-Being Index (WHO-5) at baseline, 6, 12 and 24 weeks. Primary outcomes would be the mean difference in change scores on the PHQ-9 and WHO-5 scales from baseline to 6, 12 and 24 weeks for the two study arms. Secondary outcomes include changed scores on the GAD7 scale from baseline to 6, 12 and 24 weeks for the two study arms, the dropout rates and the satisfaction rates at 12 and 24 weeks for participants in the two treatment arms. All outcome measures would be analyzed using descriptive and inferential statistics. Qualitative data will be analyzed using thematic analysis aided by NVIVO software.

Results: We expect the study results to be available within 18 months of study commencement.

Conclusion: The results of this study will shed light on the feasibility, acceptability and effectiveness of using automated email supportive message interventions in the management of patients with MDD.

DETAILED DESCRIPTION:
Depression is a debilitating condition which is characterized by changes in mood, self-attitude, cognitive functioning, sleep, appetite, and energy levels. Depression causes a decrease in quality of life that leads to impairment in occupational and social functioning. In 2010, it was estimated that mental and substance use disorders were the leading cause of years lived with disability worldwide, with Depressive disorders in particular accounting for 40·5% of disability-adjusted life-years caused by mental and substance use disorders. Depression is thus a major contributor to the overall global burden of disease and it is projected by the World Health Organization, that by 2030, Major Depressive Disorder (MDD) will be the leading cause of disability worldwide.

In 2012, over 3.2 million Canadians over 15 (11.3%) years reported symptoms of major depression and a higher health and service utilization amongst patients with depression have been reported compared to other patients. Psycho-social interventions and pharmacotherapy is the preferred first-line treatment for severe mental health problems including major depression. Psychotherapies, such as cognitive behavior therapy, interpersonal psychotherapy, problem-solving and behavioral activation are common and effective forms of treatment for depression. However, access to these psychotherapies are often limited by human resource capacity constraints and most people with depressive disorders do not receive treatment. Psychosocial services are also mostly found in cities and towns, with reduced access for rural inhabitants. Even in cities and towns these services are mostly only available during the working days and day time business hours, with caregivers often dealing with double the recommended number of clients, further restricting appointment availability. Long wait times to access counselling services and the stigma associated with seeking mental health counselling also compound the problem. In the 2012 Canadian Community Health Survey on Mental Health, barriers such as lack of readily available care system, stigma and affordability of health care services, were reported by 2.3 million Canadians who expressed they had unmet or partially met mental health care needs. It is clear, that traditional ways of providing mental healthcare alone will not be able to meet the demands for services given that the prevalence of depression is so high and not likely to decrease any time soon. There is, therefore, the need to develop innovative psychological interventions which are not human resource intensive, are easily accessible, cost-effective, are geographic location independent, scalable, and can be offered to thousands of people simultaneously.

Digital technologies for the provision of health care interventions have advanced significantly in the last decade and further development of this field looks very promising. The new technologies may enhance access to mental healthcare and contribute to closing the treatment gap that has existed over the years. Current evidence supports the efficacy and cost-effectiveness of tele mental health, especially in the context of treating depressive disorders. Useful communication methods for the delivery of mental health services includes smartphone apps, text messages and e-mails.

Supportive text messages have become an appropriate and acceptable means of delivering psychological care to patients with mental health issues. It is estimated that 99% of received mobile text messages are opened, and 90% of all text messages are read within three minutes of reception and present an opportunity to aid in the closure of the psychological treatment gap for patients with depression. In three randomized controlled trials conducted in Ireland and Canada, patients with MDD who received twice-daily supportive text messages had significantly greater reductions in their depression symptom scores compared to patients who received the usual treatment. In the first of two studies conducted in Ireland, after three months, the mean difference in change Becks Depression Inventory (BID)-II scores between the intervention and the control group was -7.9 (95% CI -13.06 to -2.76, Cohen'sd=0.85) in favor of the intervention group. Similar results were reported in another Irish study with larger sample size and in a Canadian study, a significant difference was found in the 3 months mean BDI scores between the intervention and control groups: (20.8 (SD = 11.7) vs. 24.9 (SD = 11.5), respectively, F (1, 60) = 4.83, p = 0.03, ηp2 = 0.07) with an effect size (Cohen's d) of 0.67. literature review of studies conducted on the effectiveness of text messaging as an adjunct therapy for mothers with postpartum depression living in low-income countries also reported a positive outcome and the mothers noted that they would love to receive psychological care via the text messaging. Several studies have also reported high user satisfaction of the supportive text message intervention and in one of these studies, 83% of subscribers to the Text4Mood program reported that the daily messages contributed to improving their overall mental wellbeing.

Anecdotally, some people have not been able to subscribe to supportive text messaging programs such as Text4Hope and Text4Mood because they do not have active cell phone numbers, with several individuals for whom these programs have been recommended in Addiction and Mental Health clinics in Edmonton enquiring if the messages could be sent to them via email. In the participants' satisfaction survey for the Text4Hope program, majority of respondents (64%), even though they had access to cell phones, were in favor of Email messaging for as part of their health care interventions during crisis periods.

In this technological period where faster, accessible and efficient communication medium is of outmost importance, e-mail has emerged and professionals have continued to used e-mail as a medium of communication, including communication between physicians with patients. The uniqueness of E-mail can be linked to its special characteristics, such as asynchronous communication and rapid message delivery. Electronic-therapy has been rapidly expanding in the last decades, with evidence suggesting that the provision of mental health services over the internet is both clinically efficacious and cost-effective even though its effects remain underutilized by the medical fraternity as a viable medium of communication. Given this introduction, the goal of this study is to evaluate the feasibility, comparative effectiveness and user satisfaction with daily supportive e-mail messaging as an intervention to treat patients with MDD when compared to daily supportive text messaging.

Our specific objectives include:

1. To compare the mean the difference/change in Patient Health Questionnaire (PHQ)-9 scores from baseline at 6, 12 and 24 weeks for patients with MDD receiving standard care plus daily supportive Email messages to those receiving standard care plus daily supportive text messages.
2. To compare the mean the difference/change in the WHO (Five) Well-Being Index (WHO-5) scores from baseline at 6, 12 and 24 week for patients with MDD receiving standard care plus daily supportive Email messages to those receiving standard care plus daily supportive text messages.
3. To compare the mean the difference/change in the Generalized Anxiety Disorder (GAD)-7 scale scores from baseline at 6, 12 and 24 week for patients with MDD receiving standard care plus daily supportive Email messages to those receiving standard care plus daily supportive text messages.
4. To compare the dropout and satisfaction rates between patients in the two treatment arms.
5. To explore the perspectives of beneficiaries and opt-out patients on their perceptions about the interventions

Intervention:

A research coordinator will assist participants who have provided written informed consent to enrol on either the email messaging or text messaging program by inputting their email address or phone numbers into online email messaging or text messaging applications which would be used to deliver the daily messages. Starting a day after enrollments, participants will receive either daily supportive text messages or daily supportive email messages. Both the email and text messages have the same content and have been crafted by mental health therapists, clinical psychologists, psychiatrists and mental health service users based on Cognitive Behaviour Therapy (CBT) principles. Each message would be scheduled to be delivered to participants cell phone or email address at 10 AM MT and each participant would receive the messages for 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Persons aged 18 years and over who have the capacity to provide informed consent.
2. Patients who have been assessed using structured clinical interviews for DSM 5and diagnosed with a Major Depressive Disorder.
3. Patients who have a cell phone with an active line and a functional email address and can access both E-mail messages and Text messages
4. Patients who accept willingly to be enrolled in the trial and agrees to sign the consent form

Exclusion Criteria:

1. Active psychotic disorders
2. Residing outside of regular cell phone and internet connection areas
3. Already subscribed to Text4Hope, Text4Mood, Text4Support or another supportive text messaging program.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire (PHQ)-9 scores | Baseline, 6, 12 and 24 weeks
  The Patient Health Questionnaire (PHQ) 9 is a self-administered diagnostic instrument for depression, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day).
  Minimal depression (score 0-4); Mild depression (score 5-9); Moderate depression (Score 10-14); Moderately severe depression (Score 15-19); Severe depression (score 20-27).
  We will monitor the change in this outcome measure at various intervals.
Change in the WHO (Five) Well-Being Index (WHO-5) | Baseline, 6, 12 and 24 weeks
  The World Health Organization- Five Well-Being Index (WHO-5) is a short self-reported measure of current mental wellbeing.
  Raw score: 0 represents worst possible quality of life and 25 represents best possible quality of life.
  Percentage score: 0 represents worst possible quality of life and 100 represents best possible quality of life.
  We will monitor the change in this outcome measure at various intervals.

SECONDARY OUTCOMES:
Change in the Generalized Anxiety Disorder Assessment (GAD-7) score | Baseline, 6, 12 and 24 weeks
  The Generalised Anxiety Disorder Assessment (GAD-7) is a seven-item instrument that is used to measure or assess the severity of generalised anxiety disorder (GAD). Each item asks the individual to rate the severity of his or her symptoms over the past two weeks. Response options include "not at all", "several days", "more than half the days" and "nearly every day". Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
  When used as a screening tool, further evaluation is recommended when the score is 10 or greater. We will monitor the change in this outcome measure at various intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Agyapong, MD,PhD, Principal Investigator — University of Alberta
Locations (1):
- Urgent Psychiatric Clinic, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available to the other members of the research team including Dr Ejemai Eboreime, Dr Reham Shalaby, Medard Adu
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Throughout the study duration, up to 5 years after the data is collected
Access Criteria: Involved in data collection, analyses or report writing

REFERENCES:
- [Background] Agyapong VIO. Coronavirus Disease 2019 Pandemic: Health System and Community Response to a Text Message (Text4Hope) Program Supporting Mental Health in Alberta. Disaster Med Public Health Prep. 2020 Oct;14(5):e5-e6. doi: 10.1017/dmp.2020.114. Epub 2020 Apr 22. PMID 32317038
- [Background] Agyapong VI, Ahern S, McLoughlin DM, Farren CK. Supportive text messaging for depression and comorbid alcohol use disorder: single-blind randomised trial. J Affect Disord. 2012 Dec 10;141(2-3):168-76. doi: 10.1016/j.jad.2012.02.040. Epub 2012 Mar 29. PMID 22464008
- [Background] Agyapong VIO, Juhas M, Ohinmaa A, Omeje J, Mrklas K, Suen VYM, Dursun SM, Greenshaw AJ. Randomized controlled pilot trial of supportive text messages for patients with depression. BMC Psychiatry. 2017 Aug 2;17(1):286. doi: 10.1186/s12888-017-1448-2. PMID 28768493
- [Background] Agyapong VI, Mrklas K, Juhas M, Omeje J, Ohinmaa A, Dursun SM, Greenshaw AJ. Cross-sectional survey evaluating Text4Mood: mobile health program to reduce psychological treatment gap in mental healthcare in Alberta through daily supportive text messages. BMC Psychiatry. 2016 Nov 8;16(1):378. doi: 10.1186/s12888-016-1104-2. PMID 27821096
- [Background] Agyapong VI, Milnes J, McLoughlin DM, Farren CK. Perception of patients with alcohol use disorder and comorbid depression about the usefulness of supportive text messages. Technol Health Care. 2013;21(1):31-9. doi: 10.3233/THC-120707. PMID 23358057
- [Background] Becker KD, Buckingham SL, Rith-Najarian L, Kline ER. The Common Elements of treatment engagement for clinically high-risk youth and youth with first-episode psychosis. Early Interv Psychiatry. 2016 Dec;10(6):455-467. doi: 10.1111/eip.12283. Epub 2015 Oct 20. PMID 26486257
- [Background] Berrouiguet S, Baca-Garcia E, Brandt S, Walter M, Courtet P. Fundamentals for Future Mobile-Health (mHealth): A Systematic Review of Mobile Phone and Web-Based Text Messaging in Mental Health. J Med Internet Res. 2016 Jun 10;18(6):e135. doi: 10.2196/jmir.5066. PMID 27287668
- [Background] Broom MA, Ladley AS, Rhyne EA, Halloran DR. Feasibility and Perception of Using Text Messages as an Adjunct Therapy for Low-Income, Minority Mothers With Postpartum Depression. JMIR Ment Health. 2015 Mar 16;2(1):e4. doi: 10.2196/mental.4074. eCollection 2015 Jan-Mar. PMID 26543910
- [Background] Chisholm D, Sweeny K, Sheehan P, Rasmussen B, Smit F, Cuijpers P, Saxena S. Scaling-up treatment of depression and anxiety: a global return on investment analysis. Lancet Psychiatry. 2016 May;3(5):415-24. doi: 10.1016/S2215-0366(16)30024-4. Epub 2016 Apr 12. PMID 27083119
- [Background] Garcia-Lizana F, Munoz-Mayorga I. Telemedicine for depression: a systematic review. Perspect Psychiatr Care. 2010 Apr;46(2):119-26. doi: 10.1111/j.1744-6163.2010.00247.x. PMID 20377799
- [Background] Hall AK, Cole-Lewis H, Bernhardt JM. Mobile text messaging for health: a systematic review of reviews. Annu Rev Public Health. 2015 Mar 18;36:393-415. doi: 10.1146/annurev-publhealth-031914-122855. PMID 25785892
- [Background] Iyer S, Jordan G, MacDonald K, Joober R, Malla A. Early intervention for psychosis: a Canadian perspective. J Nerv Ment Dis. 2015 May;203(5):356-64. doi: 10.1097/NMD.0000000000000288. PMID 25900548
- [Background] Kerst A, Zielasek J, Gaebel W. Smartphone applications for depression: a systematic literature review and a survey of health care professionals' attitudes towards their use in clinical practice. Eur Arch Psychiatry Clin Neurosci. 2020 Mar;270(2):139-152. doi: 10.1007/s00406-018-0974-3. Epub 2019 Jan 3. PMID 30607530
- [Background] Lal S, Malla A. Service Engagement in First-Episode Psychosis: Current Issues and Future Directions. Can J Psychiatry. 2015 Aug;60(8):341-5. doi: 10.1177/070674371506000802. PMID 26454555
- [Background] Lowe B, Kroenke K, Herzog W, Grafe K. Measuring depression outcome with a brief self-report instrument: sensitivity to change of the Patient Health Questionnaire (PHQ-9). J Affect Disord. 2004 Jul;81(1):61-6. doi: 10.1016/S0165-0327(03)00198-8. PMID 15183601
- [Background] Mohr DC, Tomasino KN, Lattie EG, Palac HL, Kwasny MJ, Weingardt K, Karr CJ, Kaiser SM, Rossom RC, Bardsley LR, Caccamo L, Stiles-Shields C, Schueller SM. IntelliCare: An Eclectic, Skills-Based App Suite for the Treatment of Depression and Anxiety. J Med Internet Res. 2017 Jan 5;19(1):e10. doi: 10.2196/jmir.6645. PMID 28057609
- [Background] Nolin M, Malla A, Tibbo P, Norman R, Abdel-Baki A. Early Intervention for Psychosis in Canada: What Is the State of Affairs? Can J Psychiatry. 2016 Mar;61(3):186-94. doi: 10.1177/0706743716632516. PMID 27254094
- [Background] Pratt LA, Brody DJ. Depression in the United States household population, 2005-2006. NCHS Data Brief. 2008 Sep;(7):1-8. PMID 19389321
- [Background] Singla DR, Raviola G, Patel V. Scaling up psychological treatments for common mental disorders: a call to action. World Psychiatry. 2018 Jun;17(2):226-227. doi: 10.1002/wps.20532. No abstract available. PMID 29856556
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Sucala M, Schnur JB, Constantino MJ, Miller SJ, Brackman EH, Montgomery GH. The therapeutic relationship in e-therapy for mental health: a systematic review. J Med Internet Res. 2012 Aug 2;14(4):e110. doi: 10.2196/jmir.2084. PMID 22858538
- [Background] Sunderland A, Findlay LC. Perceived need for mental health care in Canada: Results from the 2012 Canadian Community Health Survey-Mental Health. Health Rep. 2013 Sep;24(9):3-9. PMID 24258361
- [Background] Versluis A, Verkuil B, Spinhoven P, van der Ploeg MM, Brosschot JF. Changing Mental Health and Positive Psychological Well-Being Using Ecological Momentary Interventions: A Systematic Review and Meta-analysis. J Med Internet Res. 2016 Jun 27;18(6):e152. doi: 10.2196/jmir.5642. PMID 27349305
- [Background] Wang PS, Lane M, Olfson M, Pincus HA, Wells KB, Kessler RC. Twelve-month use of mental health services in the United States: results from the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):629-40. doi: 10.1001/archpsyc.62.6.629. PMID 15939840
- [Background] Wells KB, Stewart A, Hays RD, Burnam MA, Rogers W, Daniels M, Berry S, Greenfield S, Ware J. The functioning and well-being of depressed patients. Results from the Medical Outcomes Study. JAMA. 1989 Aug 18;262(7):914-9. PMID 2754791
- [Background] Whiteford HA, Degenhardt L, Rehm J, Baxter AJ, Ferrari AJ, Erskine HE, Charlson FJ, Norman RE, Flaxman AD, Johns N, Burstein R, Murray CJ, Vos T. Global burden of disease attributable to mental and substance use disorders: findings from the Global Burden of Disease Study 2010. Lancet. 2013 Nov 9;382(9904):1575-86. doi: 10.1016/S0140-6736(13)61611-6. Epub 2013 Aug 29. PMID 23993280
- [Background] Wu Z, Penning MJ, Schimmele CM. Immigrant status and unmet health care needs. Can J Public Health. 2005 Sep-Oct;96(5):369-73. doi: 10.1007/BF03404035. PMID 16238157
- [Background] Zhou X, Snoswell CL, Harding LE, Bambling M, Edirippulige S, Bai X, Smith AC. The Role of Telehealth in Reducing the Mental Health Burden from COVID-19. Telemed J E Health. 2020 Apr;26(4):377-379. doi: 10.1089/tmj.2020.0068. Epub 2020 Mar 23. No abstract available. PMID 32202977
- [Derived] Adu MK, Eboreime O, Shalaby R, Eboreime E, Agyapong B, da Luz Dias R, Sapara AO, Agyapong VIO. Comparing Email Versus Text Messaging as Delivery Platforms for Supporting Patients With Major Depressive Disorder: Noninferiority Randomized Controlled Trial. JMIR Form Res. 2024 Sep 9;8:e59003. doi: 10.2196/59003. PMID 39250182
- [Derived] Adu MK, Shalaby R, Eboreime E, Sapara A, Nkire N, Chawla R, Chima C, Achor M, Osiogo F, Chue P, Greenshaw AJ, Agyapong VI. Text Messaging Versus Email Messaging to Support Patients With Major Depressive Disorder: Protocol for a Randomized Hybrid Type II Effectiveness-Implementation Trial. JMIR Res Protoc. 2021 Oct 13;10(10):e29495. doi: 10.2196/29495. PMID 34643541
- See also: E-mail communication: Issues for mental health counselors — https://doi.org/10.17744/mehc.33.1.05208025375v03r7
- See also: Personalized treatment for functional outcome in depression — https://research.vu.nl/en/publications/personalized-treatment-for-functional-outcome-in-depression
- See also: The Global burden of disease : a comprehensive assessment of mortality and disability from diseases, injuries, and risk factors in 1990 and projected to 2020 : summary / edited by Christopher J. L. Murray, Alan D. Lopez — https://apps.who.int/iris/handle/10665/41864